CLINICAL TRIAL: NCT07194148
Title: Comparison of the Effectiveness of the Digital Gamification Training Method Developed for Total Hip Replacement Surgery Instrument Table Layout and the Traditional Training Method: A Randomized Controlled Trial
Brief Title: Digital Gamification vs. Traditional Training for Hip Replacement Instrument Table Setup (ORNurse)
Acronym: ORNurse
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: DERYA ESENKAYA (Other)
Responsible Party: Sponsor-Investigator, DERYA ESENKAYA, Principal Investigator, Bozok University
Organization: Bozok University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: BozokU-TKP2025-01
Record Dates: First submitted 2025-09-18; First posted 2025-09-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Surgical Education; Operating Room Nursing; Educational Technology
Keywords: Digital Gamification; Surgical Instrument Table; Nursing Education; Educational Technology

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to either the digital gamification group or the traditional training group.
Masking Description: No masking was applied since participants and researchers are aware of the assigned intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Digital Gamification Group (Experimental): Participants in this group will receive educational training using a custom-developed digital gamified simulation platform (ORNurse: Steril Setup 1.0) designed to teach surgical instrument table setup for total hip replacement surgery. Training includes interactive 3D simulation tasks and self-paced learning modules.
  Intervention:
  Name: Behavioral: Gamified Digital Education (ORNurse: Steril Setup 1.0) Other Names: ORNurse Game, Surgical Instrument Training Simulation
  Description:
  "A digital game developed to train surgical instrument table setup. Participants interact with simulation tasks and receive immediate feedback."
  Interventions: Behavioral: Gamified Digital Education (ORNurse: Steril Setup 1.0)
- Traditional Training Group (Active Comparator): Participants in this group will receive standard educational training consisting of a lecture-based presentation and printed materials on instrument table setup for total hip replacement surgery, delivered in a classroom setting.
  Intervention:
  Name: Behavioral: Traditional Training Other Names: Lecture-based Education, Printed Training Materials
  Description:
  "A classroom-based lecture accompanied by printed materials covering the correct surgical instrument table setup."
  Interventions: Behavioral: Traditional Training

INTERVENTIONS:
Behavioral: Gamified Digital Education (ORNurse: Steril Setup 1.0) — A behavioral intervention utilizing a custom-developed 3D digital game designed to teach perioperative nurses or students the correct layout of surgical instrument tables in total hip arthroplasty. The game includes interactive modules, feedback mechanisms, and simulated scenarios based on a validated protocol.
  Other Names: ORNurse Game, Surgical Instrument Training Simulation
  Arms: Digital Gamification Group
Behavioral: Traditional Training — A classroom-based lecture accompanied by printed materials covering the correct surgical instrument table setup for total hip replacement surgery.
  Other Names: Lecture-based Education; Printed Training Materials
  Arms: Traditional Training Group

SUMMARY:
This randomized controlled trial aims to compare the effectiveness of a digital gamification-based training method and a traditional training method on instrument table layout skills in total hip replacement surgery. Nursing students will be randomly assigned to either a game-based learning group or a control group receiving conventional education. The primary outcome is the accuracy of surgical instrument placement. The study will be conducted at Bozok University in Turkey.

DETAILED DESCRIPTION:
This study was designed to address the lack of standardized training protocols in instrument table setup for total hip arthroplasty. A digital gamified training tool (ORNurse: Steril Setup 1.0) was developed based on a validated surgical table protocol and integrated with a 3D simulation environment. The intervention group will receive hands-on training through the game, while the control group will receive traditional lecture-based training. The study will evaluate the effectiveness of the training methods on instrument layout accuracy, as well as participants' satisfaction and knowledge retention. This study aims to improve perioperative nursing education and promote standardization in surgical preparation processes.

ELIGIBILITY:
Inclusion Criteria:

Aged 18 years or older

Nursing students or perioperative nurses

No prior formal training in surgical instrument table setup for total hip arthroplasty

Willing and able to participate in digital or traditional training sessions

Provided informed consent

Exclusion Criteria:

Prior experience with surgical instrument table setup in orthopedic surgeries

Visual, cognitive, or motor impairments that limit ability to complete training tasks

Currently participating in another interventional education study

Refusal to participate or withdraws consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2025-12-15 (Estimated); Study Completion 2026-01-15 (Estimated)

PRIMARY OUTCOMES:
Mean score on the Total Hip Replacement Instrument Table Checklist (0-100 points; higher scores = more accurate layout) | Within 1 week after the intervention (post-training assessment)
  The standardized checklist consists of 20 items. Each item is scored as correct (5 points) or incorrect (0 points). The total score ranges from 0 to 100. Higher scores indicate more accurate placement and organization of surgical instruments on the sterile table.

SECONDARY OUTCOMES:
Mean score on the Training Satisfaction Questionnaire (5-point Likert scale; 1 = very dissatisfied, 5 = very satisfied; higher scores = greater satisfaction) | Immediately after training session
  The Training Satisfaction Questionnaire includes 10 items evaluating clarity, usability, and overall training experience. Each item is scored from 1 (very dissatisfied) to 5 (very satisfied). The mean total score is calculated, with higher scores indicating greater satisfaction with the training method.

CONTACTS AND LOCATIONS:
Overall Officials: Emine İYİGÜN, Professor, PhD, RN, Study Director — Gülhane Faculty of Nursing, University of Health Sciences
Locations (1):
- Bozok University, School of Health Services (SHMYO), Yozgat, Yozgat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) from this study with other researchers. The collected data will be used exclusively for internal analysis and reporting purposes within the scope of the principal investigator's doctoral research. No external data sharing will occur.